CLINICAL TRIAL: NCT04776863
Title: Evaluation of the Effect of Smokeless Tobacco on Anterior Segment Parameters
Brief Title: Effect of Smokeless Tobacco on Anterior Segment
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Abdullah Beyoğlu, Assist of Prof, Kahramanmaras Sutcu Imam University
Other Study IDs: decision no: 285 dated:24-2018
Record Dates: First submitted 2021-01-11; First posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Eye Manifestations; Tobacco; Use, Harmful; Tobacco Chewing Toxicity
Keywords: Optical biometry; pupillar diameter; smokeless tobacco
MeSH Terms: conditions — Eye Manifestations; Tobacco Use

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Smokeless tobacco: Individuals using smokeless tobacco
  Interventions: Device: optical biometry measurement
- No smokeless tobacco: Individuals who do not use smokeless tobacco
  Interventions: Device: optical biometry measurement

INTERVENTIONS:
Device: optical biometry measurement — The measurements of the individuals using smokeless tobacco and those who do not were taken by optical biometry.

SUMMARY:
Observational, comparative, cross-sectional study

DETAILED DESCRIPTION:
To evaluate the acute and chronic effects of smokeless tobacco (ST) on the anterior segment parameters using optical biometry. Observational, comparative, cross-sectional study Place and Duration of Study: Department of Ophthalmology, Kahramanmaras Sutcu Imam University.

The study included 53 right eyes of 53 subjects (study group), who used ST and 54 right eyes of 54 healthy subjects without ST (control group). Following a full ophthalmological examination, baseline measurements were taken with optical biometry and these measurements were repeated at 5, 30 and 60 mins after using ST.

ELIGIBILITY:
Inclusion Criteria:

* A subject who use ST
* A subject who was not using ST

Exclusion Criteria:

* Refractive disorder
* Systemic chronic disease (diabetes, hypertension, neurological, etc.)
* Ocular trauma
* Ocular surgery
* Glaucoma
* Optic disc abnormalities
* Congenital anomaly

Ages: 26 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All the study subjects underwent a full ophthalmological examination.The anterior segment parameter measurements were taken with optical biometry.
  Each subject was questioned in respect of how many years and how many times a day they used ST. Before taking the optical biometry measurements, the subjects were questioned as to whether they had used ST, drunk anything containing caffeine or smoked cigarettes in the previous 12 hours, and those who had were excluded from the study.
  Each subject was given 1mg ST and the optical biometry measurements were repeated after 5, 30 and 60 mins. A single measurement was performed with optical biometry in the control group. To avoid diurnal variations, the measurements were taken in the morning between 09.00 and 12.00 hours.
Sampling Method: Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Central Corneal Thickness (CCT) | Baseline to 60 minutes after intervention
  Change in Central Corneal Thickness (CCT
Axial Length (AL) | Baseline to 60 minutes after intervention
  Change in Axial Length (AL)
Anterior chamber deep (ACD) | Baseline to 60 minutes after intervention
  Change in Anterior chamber deep (ACD)
Lens thickness (LT) | Baseline to 60 minutes after intervention
  Change in Lens thickness (LT)
Pupillary diameter (PD) | Baseline to 60 minutes after intervention
  Change in Pupillary diameter (PD)

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Beyoğlu, Study Chair — Kahramanmaras Sutcu Imam University
Locations (1):
- Abdullah Beyoğlu, Kahramanmaraş, None Selected, Turkey (Türkiye)